CLINICAL TRIAL: NCT02760017
Title: Evaluation of Clinical Efficacy Capsules Containing Standardized Extract of Bauhinia Forficata (Pata- De-vaca) in Diabetic Patients
Brief Title: Bauhinia Forficata in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Felipe Dal Pizzol, MD, PhD, Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 401336/2013-1
Record Dates: First submitted 2016-04-28; First posted 2016-05-03 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): capsules containing placebo for B forticata
  Interventions: Drug: Placebo
- B. forficata (Experimental): capsules of B. forficata containing 200 mg of plant extracts
  Interventions: Drug: B. forficata

INTERVENTIONS:
Drug: B. forficata
  Arms: B. forficata
Drug: Placebo
  Arms: placebo

SUMMARY:
Among the plants most used in folk medicine for the treatment of diabetes are the species of the genus Bauhinia (Fabaceae), popularly known in Brazil as "pata-de-vaca". Of these, Bauhinia forficata has the highest number of studies regarding the hypoglycemic activity. Due to this fact it is included in the Medicinal Plants List of the Brazilian Public Health System. Extracts of pata-de-vaca (B. forficata) have been explored both in relation to its chemical composition and its pharmacological potential. From the chemical point of view the main components identified in hydro alcoholic extract of the leaves are O-glycosylated derivatives of kaempferol and quercetin. Regarding pharmacological properties preclinical studies have confirmed the hypoglycemic effect and antidiabetic of the hydroalcoholic extract of the leaves of B. forficata. The search for evidence of the alleged anti-diabetic activity of B. forficata in clinical level was performed in only two studies, both with few patients, and questionable methodological quality that used tea as a pharmaceutical form, a fact that allows us to question the validity of data considering the risks of no dose reproducibility ingested by patients during the study. Thus the investigators here intend to determine the effects of a standardized extract of B. forficata in the control of patients with diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetic patients
* Using oral antidiabetic treatment for at least 3 months
* Glycated hemoglobin levels > 7.5% or
* Fasting glucose levels >=100mg/dl

Exclusion Criteria:

* Type 1 diabetes patients
* History of cancer under treatment
* Major cardiovascular event during the last 90 days (eg. stroke, myocardial infarction)
* Pregnancy
* Lactation
* Serious diseases presenting limited short-term prognosis (eg stage IV COPD end-stage heart failure)
* Child B or C cirrhotic patients
* Patients with chronic renal failure on dialysis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
glycated hemoglobin levels | 4 months
fasting glucose levels | 4 months

SECONDARY OUTCOMES:
Plasma inflammatory parameters levels | 4 months
  Interleukin-6 and c-reactive protein levels
Plasma oxidative stress parameters levels | 4 months
  Advanded glycation end-products, protein carbonyl and lipid peroxidation levels
Plasma endothelin-1 levels | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade do Extremo Sul Catarinense, Criciúma, Santa Catarina, Brazil